CLINICAL TRIAL: NCT03643952
Title: A Phase II Open-Label, Single-arm Clinical Trial to Study the Safety, Efficacy and Pharmacokinetics of MK-3009 (Daptomycin) in Japanese Pediatric Participants Aged 1 to 17 Years With Complicated Skin and Soft Tissue Infections or Bacteremia Caused by Gram-positive Cocci
Brief Title: Safety, Efficacy, and Pharmacokinetics (PK) of Daptomycin (MK-3009) in Japanese Pediatric Subjects With Complicated Skin and Soft Tissue Infections (cSSTI) and Bacteremia (MK-3009-029)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3009-029; MK-3009-029 (Other: Merck Protocol Number); 184155 (Registry Identifier: JAPIC-CTI); 2020-001576-15 (EudraCT Number)
Record Dates: First submitted 2018-08-21; First posted 2018-08-23 (Actual); Results first posted 2021-03-30 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-04

CONDITIONS: Bacteremia; Soft Tissue Infections; Skin Diseases, Infectious
Keywords: methicillin-resistant S. aureus (MRSA) infections; complicated skin and soft tissue infections (cSSTI)
MeSH Terms: conditions — Bacteremia; Soft Tissue Infections; Skin Diseases, Infectious; Infections | interventions — Daptomycin; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daptomycin (Experimental): Participants aged 1 to 17 years old with cSSTI or bacteremia will receive daptomycin intravenously every 24 hours for either 5-14 days for cSSTI or for 5-42 days for bacteremia.
  Interventions: Drug: Daptomycin for Injection

INTERVENTIONS:
Drug: Daptomycin for Injection — Once daily administration of 5, 7, 9, 10, or 12 mg/kg intravenous (IV) daptomycin infused with 25-50 mL saline over 30-60 minutes depending upon infection type and age level.
  Other Names: MK-3009

SUMMARY:
The purpose of this study is to assess the safety, efficacy and pharmacokinetic (PK) parameters of daptomycin for injection in Japanese pediatric participants aged 1 to 17 years with complicated skin and soft tissue infection (cSSTI) or bacteremia caused by gram-positive cocci.

ELIGIBILITY:
Inclusion Criteria:

* Requires treatment for cSSTI or bacteremia.
* Is male or female Japanese aged ≥ 1 to ≤ 17 years on the day of signing informed consent.
* As a male participant, has agreed to use contraception during the treatment period and for at least 14 days after the last dose of study treatment and refrain from donating sperm during this period.
* As a female participant, has agreed to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: not a woman of childbearing potential (WOCBP) or a WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 14 days after the last dose of study treatment.
* Has agreed to allow any bacterial isolates obtained from protocol-required specimens related to the current infection to be provided the Central Microbiology Reference Laboratory for study-related microbiological testing, long-term storage, and other future testing.

cSSTI Participants

* Has cSSTI known or suspected to be caused by gram-positive cocci that requires intravenous antibiotic treatment and diagnosed with either Gram stain or culture.
* Has at least 3 of the following clinical signs and symptoms associated with the cSSTI: pain, tenderness to palpation, temperature >37.0°C axillary or >37.5°C oral or >38.0° C rectal, forehead, or aural, white blood count (WBC) >12,000/mm^3 or ≥10% bands, swelling and/or induration, erythema (>1 cm beyond edge of wound or abscess), pus formation, CRP > upper limited of normal.

Bacteremia Participants

* Have proven bacteremia with pathogen identification of gram-positive cocci at least one blood culture bottle by conventional culture methods or by a rapid diagnostic test in screening period.
* Have probable bacteremia with a blood culture result demonstrating gram-positive cocci by Gram stain in screening period.

Exclusion Criteria:

* Has received previous systemic antimicrobial therapy that is effective against gram-positive cocci and exceeding 72 hours duration administered at any time during the 96 hours prior to the first dose of study drug.
* Has a known infection caused solely by gram-negative pathogen(s), fungus(i) or virus(es).
* Has pneumonia (septic emboli in the lung is not an exclusion if clear evidence of source of infection is other than lungs), empyema, meningitis, endocarditis, or osteoarticular infection.
* Has a history of or current rhabdomyolysis.
* Is anticipated to require non-study systemic antibiotics that may be potentially effective against gram-positive pathogen(s).
* Has shock or hypotension unresponsive to fluids or vasopressors for ≥ 4 hours.
* Has significant allergy/hypersensitivity or intolerance to daptomycin.
* Has renal insufficiency.
* Has a history of clinically significant (as assessed by the Investigator) muscular disease, nervous system or seizure disorder, including unexplained muscular weakness, history of peripheral neuropathy, Guillain-Barre or spinal cord injury; previous uncomplicated febrile seizure allowed.
* Has a history or current evidence of any condition, therapy, lab abnormality or other circumstance that might expose the participant to risk by participating in the trial, confound the results of the trial, or interfere with the participant's participation for the full duration of the trial.
* Is a female who is pregnant or is expecting to conceive (or is a male partner of a female who is expecting to conceive), is breastfeeding, or plans to breastfeed prior to completion of the study.
* Is currently participating in, or has participated in, any other clinical study involving the administration of investigational or experimental medication (not licensed by regulatory agencies) at the time of the presentation or during the previous 30 days prior to screening or is anticipated to participate in such a clinical study during the course of this trial.
* Has previously participated in this study at any time.
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is investigational site or sponsor staff directly involved with this study.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (16):
- Japan (16):
  - Japan Community Health Care Organization Chukyo Hospital ( Site 0030), Nagoya, Aichi-ken
  - Japan Community Health care Organization Kyushu Hospital ( Site 0016), Kitakyushu, Fukuoka
  - Maebashi Red Cross Hospital ( Site 0012), Maebashi, Gunma
  - Kobe University Hospital ( Site 0015), Kobe, Hyōgo
  - Shikoku Medical Center for Children and Adults ( Site 0027), Zentsujichó, Kagawa-ken
  - Showa University Fujigaoka Hospital ( Site 0023), Yokohama, Kanagawa
  - Kanagawa Children's Medical Center ( Site 0025), Yokohama, Kanagawa
  - National Hospital Organization National Mie Hospital ( Site 0002), Tsu, Mie-ken
  - National Hospital Organization Beppu Medical Center ( Site 0003), Beppu, Oita Prefecture
  - Tokyo Metropolitan Children's Medical Center ( Site 0004), Fuchū, Tokyo
  - Chiba University Hospital ( Site 0005), Chiba
  - Chiba Children's Hospital ( Site 0024), Chiba
  - National Hospital Organization Kumamoto Medical Center ( Site 0018), Kumamoto
  - Osaka City General Hospital ( Site 0020), Osaka
  - Saitama City Hospital ( Site 0008), Saitama
  - Nihon University Itabashi Hospital ( Site 0029), Tokyo

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Iwata S, Koyama H, Murata Y. Efficacy and safety of daptomycin in Japanese pediatric participants with complicated skin and soft tissue infections or bacteremia caused by gram-positive cocci. J Infect Chemother. 2022 Mar;28(3):406-412. doi: 10.1016/j.jiac.2021.11.019. Epub 2021 Dec 15. PMID 34920946

RESULTS

PARTICIPANT FLOW:
Groups:
- Daptomycin: Participants aged 1 to 17 years old with complicated skin and soft tissue infections (cSSTI) or bacteremia received daptomycin intravenously every 24 hours for either 5-14 days for cSSTI or for 5-42 days for bacteremia.
Period: Overall Study
Arm/Group | Daptomycin
Started | 18
Completed | 17
Not Completed | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Groups:
- Daptomycin: Participants aged 1 to 17 years old with cSSTI or bacteremia received daptomycin intravenously every 24 hours for either 5-14 days for cSSTI or for 5-42 days for bacteremia.
Arm/Group | Daptomycin
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 6.9 (5.1)
Age, Customized [Number; unit: Participants]
  Newborns (0-27 days) | 0
  Infants and toddlers (28 days-23 months) | 5
  Children (2-11 years) | 9
  Adolescents (12-17 years) | 4
  Adults (18-64 years) | 0
  From 65-84 years | 0
  85 years and over | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 18
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Adverse Event
Description: An adverse event (AE) is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an adverse event.
Time Frame: Up to 56 days
Population: All enrolled participants who received at least one dose of daptomycin
Measure: Number; unit: Percentage of Participants
Arm/Group | Daptomycin
Number analyzed (Participants) | 18
Percentage of Participants | 55.6

2. Primary Outcome: Percentage of Participants That Discontinued Study Treatment Due to an Adverse Event (AE)
Description: An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an adverse event.
Time Frame: Up to 42 days
Population: All enrolled participants who received at least one dose of daptomycin
Measure: Number; unit: Percentage of Participants
Arm/Group | Daptomycin
Number analyzed (Participants) | 18
Percentage of Participants | 0

3. Secondary Outcome: Percentage of Participants With Methicillin-Resistant Staphylococcus Aureus (MRSA) Infections Who Experienced Clinical Success
Description: Clinical success in participants with MRSA infections was defined as either "Cure" - Resolution of clinically significant signs and symptoms associated with admission infection and no further antibiotic therapy required, OR "Improved"- partial resolution of clinical signs or symptoms of infection with no further antibiotic therapy required.
Time Frame: Up to 7 days following end of treatment (up to 49 days)
Population: All enrolled participants with cSSTI or bacteremia who had a positive culture of MRSA at baseline and received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Daptomycin (MRSA With cSSTI): Participants aged 1 to 17 years old with cSSTI and a positive culture of MRSA at baseline received daptomycin intravenously every 24 hours for 5-14 days.
- Daptomycin (MRSA With Bacteremia): Participants aged 1 to 17 years old with bacteremia and a positive culture of MRSA at baseline received daptomycin intravenously every 24 hours for 5-42 days.
Arm/Group | Daptomycin (MRSA With cSSTI) | Daptomycin (MRSA With Bacteremia)
Number analyzed (Participants) | 7 | 1
Percentage of Participants | 85.7 [42.1 to 99.6] | 100 [2.5 to 100]

4. Secondary Outcome: Percentage of Participants With MRSA Infections Who Experienced a Microbiological Response
Description: Participant-level microbiological response in participants with MRSA infections at baseline is defined as absence or presumed absence of all baseline infecting pathogens AND no gram-positive superinfection or gram-positive new infection, as assessed by infection site specimen culture or blood culture.
Time Frame: Up to 7 days following end of treatment (up to 49 days)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Daptomycin (MRSA With cSSTI) | Daptomycin (MRSA With Bacteremia)
Number analyzed (Participants) | 7 | 1
Percentage of Participants | 71.4 [29.0 to 96.3] | 100 [2.5 to 100]

5. Secondary Outcome: Area Under the Concentration Time Curve From 0 to 24 Hours (AUC0-24hr) of Daptomycin
Description: Blood samples were collected at pre-specified time points to determine the AUC0-24 of daptomycin.
Time Frame: Pre-dose and at 15 minutes, 1 hour, 4 hours, and 12 hours post-dose on Day 3 of daptomycin treatment
Population: All enrolled participants who received at least 3 consecutive intravenous (IV) infusions of study treatment, had at least 1 pharmacokinetic (PK) sample following study drug administration, and did not have any protocol violations affecting the PK profile
Measure: Mean (Standard Deviation); unit: µg·hr/mL
Groups:
- Daptomycin (cSSTI): Participants with cSSTI received daptomycin intravenously every 24 hours for 5-14 days.
- Daptomycin (Bacteremia): Participants with bacteremia received daptomycin intravenously every 24 hours for 5-42 days.
Arm/Group | Daptomycin (cSSTI) | Daptomycin (Bacteremia)
Number analyzed (Participants) | 14 | 3
µg·hr/mL
  Age Category 1-<2 years: number analyzed (Participants) | 3 | 1
  Age Category 1-<2 years | 574 (99.1) | 502 (0)
  Age Category 2-6 years: number analyzed (Participants) | 3 | 0
  Age Category 2-6 years | 431 (53.6) |
  Age Category 7-11 years: number analyzed (Participants) | 5 | 1
  Age Category 7-11 years | 409 (143) | 599 (0)
  Age Category 12-17 years: number analyzed (Participants) | 3 | 1
  Age Category 12-17 years | 316 (18.2) | 422 (0)

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Daptomycin
Description: Blood samples were collected at pre-specified timepoints to determine Cmax of daptomycin.
Time Frame: Pre-dose and at 15 minutes, 1 hour, 4 hours, and 12 hours post-dose on Day 3 of daptomycin treatment
Population: All enrolled participants who received at least 3 consecutive IV infusions of study treatment, had at least 1 PK sample following study drug administration, and did not have any protocol violations affecting the PK profile
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- Daptomycin (cSSTI): Participants diagnosed with cSSTI received daptomycin intravenously every 24 hours for 5-14 days.
Arm/Group | Daptomycin (cSSTI) | Daptomycin (Bacteremia)
Number analyzed (Participants) | 14 | 4
μg/mL
  Age Category 1-<2 years: number analyzed (Participants) | 3 | 2
  Age Category 1-<2 years | 91.7 (6.66) | 104 (8.70)
  Age Category 2-6 years: number analyzed (Participants) | 3 | 0
  Age Category 2-6 years | 80.3 (4.48) |
  Age Category 7-11 years: number analyzed (Participants) | 5 | 1
  Age Category 7-11 years | 64.4 (15.1) | 73.1 (0)
  Age Category 12-17 years: number analyzed (Participants) | 3 | 1
  Age Category 12-17 years | 49.3 (1.33) | 94.0 (0)

7. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Daptomycin
Description: Blood samples were collected at pre-specified time points to determine Tmax of daptomycin
Time Frame: Pre-dose and at 15 minutes, 1 hour, 4 hours, and 12 hours post-dose on Day 3 of daptomycin treatment
Population: as for outcome 6
Measure: Median (Full Range); unit: Hours
Arm/Group | Daptomycin (cSSTI) | Daptomycin (Bacteremia)
Number analyzed (Participants) | 14 | 4
Hours
  Age Category 1-<2 Years: number analyzed (Participants) | 3 | 2
  Age Category 1-<2 Years | 1.33 [1.33 to 1.37] | 1.27 [1.20 to 1.33]
  Age Category 2-6 Years: number analyzed (Participants) | 3 | 0
  Age Category 2-6 Years | 1.23 [1.12 to 1.27] |
  Age Category 7-11 Years: number analyzed (Participants) | 5 | 1
  Age Category 7-11 Years | 0.833 [0.783 to 1.00] | 0.800 [0.800 to 0.800]
  Age Category 12-17 Years: number analyzed (Participants) | 3 | 1
  Age Category 12-17 Years | 0.750 [0.750 to 0.750] | 0.733 [0.733 to 0.733]

8. Secondary Outcome: Body Weight Adjusted Clearance (CLss/wt) of Daptomycin
Description: Blood samples were collected at pre-specified time points to determine CLss/wt of daptomycin at steady state.
Time Frame: Pre-dose and at 15 minutes, 1 hour, 4 hours, and 12 hours post-dose on Day 3 of daptomycin treatment
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mL/hr/kg
Arm/Group | Daptomycin (cSSTI) | Daptomycin (Bacteremia)
Number analyzed (Participants) | 14 | 3
mL/hr/kg
  Age Category 1-<2 Years: number analyzed (Participants) | 3 | 1
  Age Category 1-<2 Years | 17.8 (2.86) | 23.9 (0)
  Age Category 2-6 Years: number analyzed (Participants) | 3 | 0
  Age Category 2-6 Years | 21.1 (2.69) |
  Age Category 7-11 Years: number analyzed (Participants) | 5 | 1
  Age Category 7-11 Years | 19.4 (8.27) | 15.0 (0)
  Age Category 12-17 Years: number analyzed (Participants) | 3 | 1
  Age Category 12-17 Years | 15.8 (0.917) | 16.6 (0)

9. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Daptomycin
Description: Blood samples were collected at pre-specified time points to determine Vss (mL) of daptomycin.
Time Frame: Pre-dose and at 15 minutes, 1 hour, 4 hours, and 12 hours post-dose on Day 3 of daptomycin treatment
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Daptomycin (cSSTI) | Daptomycin (Bacteremia)
Number analyzed (Participants) | 14 | 3
mL
  Age Category 1-<2 Years: number analyzed (Participants) | 3 | 1
  Age Category 1-<2 Years | 1146 (299) | 1918 (0)
  Age Category 2-6 Years: number analyzed (Participants) | 3 | 0
  Age Category 2-6 Years | 1753 (486) |
  Age Category 7-11 Years: number analyzed (Participants) | 5 | 1
  Age Category 7-11 Years | 3929 (2032) | 4013 (0)
  Age Category 12-17 Years: number analyzed (Participants) | 3 | 1
  Age Category 12-17 Years | 6414 (1086) | 5106 (0)

10. Secondary Outcome: Apparent Terminal Half-Life (t½) of Daptomycin
Description: Blood samples were collected at pre-specified time points to determine the t½ of daptomycin.
Time Frame: Pre-dose and at 15 minutes, 1 hour, 4 hours, and 12 hours post-dose on Day 3 of daptomycin treatment
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Hours
Groups:
- Daptomycin (Bacterermia): Participants with bacteremia received daptomycin intravenously every 24 hours for 5-42 days.
Arm/Group | Daptomycin (cSSTI) | Daptomycin (Bacterermia)
Number analyzed (Participants) | 14 | 3
Hours
  Age Category 1-<2 Years: number analyzed (Participants) | 3 | 1
  Age Category 1-<2 Years | 4.94 (0.460) | 4.46 (0)
  Age Category 2-6 Years: number analyzed (Participants) | 3 | 0
  Age Category 2-6 Years | 3.87 (0.514) |
  Age Category 7-11 Years: number analyzed (Participants) | 5 | 1
  Age Category 7-11 Years | 5.07 (1.09) | 5.85 (0)
  Age Category 12-17 Years: number analyzed (Participants) | 3 | 1
  Age Category 12-17 Years | 5.71 (0.942) | 3.98 (0)

ADVERSE EVENTS:
Time Frame: Up to 56 days
Description: All enrolled participants who received at least one dose of daptomycin
Arm/Group | Daptomycin
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 10/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daptomycin (N=18)
Constipation (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal mucosal disorder (Gastrointestinal disorders) | 1 (1)
Catheter site related reaction (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Infusion site swelling (General disorders) | 1 (1)
Injection site pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Genital candidiasis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Platelet count increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was concluded due to the difficulty of enrolling pediatric patients into the study during the COVID-19 pandemic. This study concluded enrollment with 18 participants, versus the 20 that were originally planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the sponsor, the investigator agrees to submit all manuscripts or abstracts to the sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT03643952/Prot_SAP_000.pdf